CLINICAL TRIAL: NCT01987674
Title: Impact of a Pre-meal Protein Drink on Metabolic Markers and Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Pre-meal Protein Drink Improve Glycemic Regulation
Acronym: PMB/T2D
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Test products expired.
Sponsor: Lund University (Other)
Collaborators: Landstinget i Kalmar Län (Other)
Responsible Party: Principal Investigator, Elin Östman, Associate professor, Lund University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dnr2013/239-31PMB
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-meal protein drink (Experimental): A dose of 100 ml is taken just before breakfast, lunch and dinner.
  Interventions: Dietary Supplement: Pre-meal protein drink
- Water drink (Placebo Comparator): A dose of 100 ml is taken just before breakfast, lunch and dinner.
  Interventions: Other: Water drink

INTERVENTIONS:
Dietary Supplement: Pre-meal protein drink
  Arms: Pre-meal protein drink
Other: Water drink
  Arms: Water drink

SUMMARY:
The purpose of this study is to investigate if a pre-meal drink containing proteins can positively influence glycaemic control in patients with type 2 diabetes mellitus. Comparison with a placebo is included.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed type 2 diabetes mellitus according to WHO criteria (1999)
* age between 30-80 years
* non well controlled diabetes with HbA1c-levels above 62 mmol/mol

Exclusion Criteria:

* pregnant or risk of becoming pregnant
* severe disease
* psychological disease, dementia or mental disability that makes it impossible to retrieve informed consent of participation
* liver disease
* kidney malfunction (GFR <60 or aspartate transaminase (ASAT)/alanine transaminase (ALT) two times higher than the normal interval

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  Glycated hemoglobin

SECONDARY OUTCOMES:
Postprandial glycemia | 16 weeks
  Meal challenge given at start and end of study with repeated blood glucose sampling over 2h.

OTHER OUTCOMES:
Homeostasis model assessment of insulin resistance (HOMA-IR) | 16 weeks
  HOMA-IR is a mathematical modelling of insulin resistance using fasting values of blood glucose and serum insulin.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindsdals hälsocentral, Kalmar, Sweden